CLINICAL TRIAL: NCT06937580
Title: Enhancing the Survival of Low Birth Weight Infants in Low Resource Settings Using an Implementation Science Approach
Brief Title: Enhancing the Survival of Low Birth Weight Infants in Low-Resource Settings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Center for Learning and Childhood Development Ghana (Unknown); Korle-Bu Teaching Hospital, Accra, Ghana (Other); Sunyani Teaching Hospital, Sunyani, Ghana (Unknown)
Responsible Party: Principal Investigator, Mufaro Kanyangarara, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00137641; 1R21HD116063-01 (NIH)
Record Dates: First submitted 2025-03-17; First posted 2025-04-22 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Low Birthweight; Preterm; Kangaroo Mother Care
Keywords: Low birthweight; Preterm; Low-resource; Kangaroo Mother Care
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: The study consists of a two-arm, unblinded individual randomized controlled trial to determine the effectiveness of receiving peer support and a Baby Box. The mothers in the intervention arm will receive the peer support and Baby Box, while the control arm will consist of mothers receiving standard care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): Peer Support and Baby Box
  Interventions: Behavioral: Peer Support and Baby Box
- Arm 2 (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: Peer Support and Baby Box — The intervention consists of five one-on-one peer support sessions and a Baby Box consisting of a woolen hat and socks for infant warmth, a cloth wrap to position the baby securely for skin-to-skin contact and improve comfort, a bar of soap for hygiene, and a real-time continuous temperature monitoring device for hypothermia detection
  Arms: Arm 1

SUMMARY:
Kangaroo Care, which includes skin-to-skin contact, exclusive breastfeeding, and timely follow-up, is a proven method to reduce neonatal morbidity and mortality in low-resource settings where the risks of prematurity, neonatal hypothermia, and neonatal mortality are high. However, numerous challenges such as inadequate knowledge, financial constraints, cultural norms, stigma, and limited social support impede its effective practice among mothers of low birthweight infants. To address these barriers, the intervention consists of informational, emotional and motivational support from trained peers and a box with warmth-related items to support the adoption and sustainment of Kangaroo Care at home. The investigators will enroll 328 mothers of low birthweight infants, who intend to initiate Kangaroo Care at two tertiary hospitals in Ghana, in a prospective randomized controlled trial. The trial aims to evaluate the effectiveness of the intervention in increasing exclusive breastfeeding rates and the duration of skin-to-skin contact at 7 and 28 days post-hospital discharge. Mothers in the control group will receive the standard of care, which consists of one counseling session on Kangaroo Care before discharge and a follow-up phone call after discharge. In addition to the standard of care, mothers in the intervention group will receive five one-on-one peer support sessions over one month, along with a box containing a hat, socks, a specialized wrap to support skin-to-skin contact, soap for hand hygiene, and a temperature monitoring device that alerts mothers if their infant becomes hypothermic. Using surveys, outcome data will be collected from both study groups at enrollment in the hospital, and at 7 and 28 days after discharge at participants' homes. Additionally, in-depth interviews will be conducted with 10-15 mothers from the intervention group, 10-15 healthcare workers, and all six peer supporters delivering the intervention. These interviews will explore the implementation of the intervention and contextualize barriers and facilitators from the perspectives of different stakeholders.

DETAILED DESCRIPTION:
Globally, about 20 million infants are born with low birthweight (LBW), and these infants face a myriad of health challenges, including difficulties in regulating body temperature, poor nutritional status, increased vulnerability to infections, and delayed development, placing emotional and financial burdens on families. Kangaroo Care (KC), consisting of continuous skin-to-skin contact, exclusive breastfeeding, and early discharge, is an evidence-based intervention recommended for LBW newborns to improve their survival and healthy development, especially in low-resource settings where the risks of prematurity, neonatal hypothermia, and neonatal mortality are disproportionately high. Despite the effectiveness of KC, widespread scale-up has been slow due to barriers to implementation and adoption. Existing efforts have primarily focused on health systems and policy changes, neglecting the need to support mothers and families to continue practicing KC at home. Several sociocultural and economic factors, including lack of essential warmth-related items, cultural norms, stigma, and limited social support, hinder the KC continuation at home. To address these challenges, an intervention grounded in the Information, Motivation, and Behavior (IMB) model has been developed. The intervention offers emotional, informational, and motivational peer support to mothers of LBW infants and a kit containing low-cost, locally sourced neonatal care items to facilitate skin-to-skin contact and breastfeeding. A type II hybrid effectiveness-implementation study will be conducted. First, the effectiveness of the intervention will be tested using an individual randomized controlled trial, enrolling 328 mother-infant dyads eligible for KC from two tertiary hospitals in Ghana (Aim 1). It is hypothesized that mothers receiving the intervention will be more likely to continue KC at home 7 days after discharge compared to those in the control group receiving the standard of care. The primary effectiveness outcome is any duration of skin-to-skin contact and exclusive breastfeeding at 7 and 28 days post-discharge. Second, the implementation process including associated barriers and facilitators to implementation will be explored using mixed methods (Aim 2). In-depth interviews will be conducted with participants, peer supporters and healthcare workers. Thematic analysis of the interviews will be guided by the Consolidated Framework for Implementation Research (CFIR) framework and combine both inductive and deductive approaches. Findings from this research will inform the development of effective models for KC implementation and scale-up.

ELIGIBILITY:
The study will consider mother-infant dyads eligible for participation if they meet all of the following criteria:

* Mothers aged between 15 and 49 years.
* Mothers intending to initiate facility-based Kangaroo Care, irrespective of gestational age, delivery mode, or singleton or multiple birth status.
* Mothers capable of providing consent or those unwilling to provide consent.
* Mothers without medical complications hindering Kangaroo Care.
* Mothers residing within a 10-kilometer radius of the study site.
* Infants capable of spontaneous breathing within 1 hour of birth.
* Infants without major congenital malformations.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Mother-infant
Enrollment: 328 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration of skin-to-skin contact based on self-report | 7 and 28 days
  Duration of skin-to-skin contact in hours and minutes will be assessed at 7 and 28 days using an interviewer-administered questionnaire to mothers.
Exclusive breastfeeding based on self-report | 7 and 28 days
  Current feeding practices will be assessed at 7 and 28 days using an interviewer-administered questionnaire to mothers.

SECONDARY OUTCOMES:
Maternal Self-Efficacy as assessed by the Perceived Maternal Parenting Self-Efficacy Tool | 7 and 28 days
  The Perceived Maternal Parenting Self-Efficacy (PMP S-E) tool is a validated 18 item scale designed to assess maternal self-efficacy in caring for preterm infants, particularly in within a hospital setting. The scale evaluates a mother's confidence in her ability to care for her newborn across various domains such as recognizing and interpreting infant cues, providing physical care, and managing emotional responses. Each item is typically rated on a 4-point Likert scale, with total scores ranging from 20 to 80. Higher scores indicate a stronger sense of maternal competence and confidence in parenting skills.
Low birthweight stigma as assessed by the Small Baby Internalized Stigma Scale (SBISS) | 7 and 28 days
  The Small Baby Internalized Stigma Scale (SBISS) is an 8 item tool to assess both internalized and externalized stigma experienced by mothers of low birthweight infants. This scale captures experiences such as shame, blame, judgment from others, and self-stigmatization. Respondents rate items on a Likert scale, typically from 1 (Strongly Disagree) to 5 (Strongly Agree), resulting in a possible score range of 8 to 40. Higher scores indicate more intense experiences of stigma and potential emotional distress related to their infant's condition.
Maternal Stress as assessed by the Perceived Stress Scale | 7 and 28 days
  The Perceived Stress Scale (PSS) is a widely used, validated 10-item scale for measuring the perception of stress within the previous month. The PSS is applicable in various populations, including postpartum mothers, where it helps assess the emotional strain associated with caregiving and life transitions. Each item is rated on a 5-point scale from 0 (Never) to 4 (Very Often), yielding total scores ranging from 0 to 40. Higher scores indicate a higher perception of stress.
Social Support as assessed by the Perinatal Infant Care Social Support Scale | 7 and 28 days
  The Perinatal Infant Care Social Support Scale (PICSS) is a 24-item measure of perceived adequacy and availability of social support from family, friends and significant others during the perinatal period. This tool evaluates the emotional, informational, and instrumental support received from family, friends, and other social connections regarding infant care. Each item is scored on a scale of 0 (Not at all helpful) to 3 (Very helpful), resulting in a total score range of 0 to 96. Higher scores indicate stronger perceived support networks and resources available to the mother during a critical developmental and emotional time.
Maternal Depression as assessed by the Edinburg Postnatal Depression Scale | 7 and 28 days
  Edinburg Postnatal Depression Scale (EPDS) is a 10-item self-report questionnaire developed to screen for symptoms of postnatal depression, especially in low-resource settings. It focuses on the emotional and psychological well-being of mothers over the previous seven days, addressing symptoms such as sadness, guilt, anxiety, and thoughts of self-harm. Each item is scored from 0 to 3, leading to a total score between 0 and 30. Higher scores indicate more severe depressive symptoms levels.
Implementation barriers and facilitators as assessed by qualitative interviews | baseline, 7 and 28 days
  In-depth interviews (IDIs) will be conducted with mothers in the intervention group, peer supporters, study nurses, and healthcare workers to evaluate intervention implementation and contextualize barriers and facilitators for implementation from the perspectives of different stakeholders. Analysis will be guided by the Consolidated Framework for Implementation Research (CFIR).

CONTACTS AND LOCATIONS:
Locations (2):
- Ghana (2):
  - Korle-Bu Teaching Hospital, Accra, Greater Accra Region
  - Sunyani Regional Teaching Hospital, Sunyani

IPD SHARING:
Plan to Share IPD: Yes
Shared data will be de-identified, and the original data will be retained at the investigator's institution. Data and metadata from this project will be archived at the Inter-university Consortium for Political and Social Research (ICPSR).
Supporting Information: Study Protocol, SAP
Time Frame: The investigators will liaise with ICPSR to allow for about 3 months before the required release date to account for any potential lag time between submission and data release. The permanently archived data will be available to domain specialists, ensuring data longevity across changing technologies, new media, and data formats.
Access Criteria: The investigators will provide analytic code for linking, merging, or manipulating datasets, which ICPSR will make available alongside the data. ICPSR will produce standardized project-level and variable-level metadata that conform to the Data Documentation Initiative (DDI) metadata standard, ensuring compatibility with other data archive catalogs. The archived data will be available for long-term access by domain specialists. Public data users will access the de-identified data through ICPSR after registration and compliance with ICPSR's Terms of Use. Data users will be bound by the Restricted Data Use Agreement, ensuring the confidentiality of human subjects.